CLINICAL TRIAL: NCT04040699
Title: A Phase Ib Study to Evaluate Efficacy, Safety and Tolerability of KN026 Combined With KN046 in Subjects With HER2 Positive Solid Tumor
Brief Title: KN026 Combined With KN046 in Subjects With HER2 Positive Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Principal Investigator, Shen Lin, MD,Professor,Chief of Department of GI Oncology,Peking University Cancer Hospital, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KN046-IST-02
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: HER2 Positive Solid Tumor
Keywords: KN026; KN046; HER2 Positive Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KN026 combined with KN046 (Experimental): KN026 is an anti-HER2 bispecific antibody that can simultaneously bind two non-overlapping epitopes of HER2, leading to a dual HER2 signal blockade.
  KN046 is a PD-L1 - CTLA-4 bispecific antibody.
  Interventions: Biological: KN026 combined with KN046

INTERVENTIONS:
Biological: KN026 combined with KN046 — KN026 and KN046 are given at 20mg/Kg and 3mg/Kg intravenously on day 1of each 2 weeks cycle at the beginning respectively.The dosage will be escalated if adverse events are tolerated according to the scheme.

SUMMARY:
This is a phase Ib, open-label, dose-escalation and expansion study to evaluate the safety, tolerability, pharmacokinetics and anti-tumor activity of KN026 combined with KN046 in subjects with advanced HER2 positive solid tumors.

DETAILED DESCRIPTION:
The study is composed of 2 stages. Stage 1 consists of dose escalation cohorts for determining the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D). Part 2 consists of 4 tumor type expansion cohorts for expanding the information on clinical safety, clinical pharmacokinetics and antitumor activity in HER2 positive patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed inform consent form (ICF)
* Age ≥ 18 years and ≤ 75 years, male or female
* Histologically or cytologically documented advanced HER2 positive solid tumor
* Received at least one prior standard therapy
* At least one measurable lesion according to Response Evaluation Criteria In Solid Tumors（RECISIT） v 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ function
* LVEF≥ 50% (ECHO)
* Female patients and males with partners of childbearing potential should be using highly effective contraceptive measures (failure rate of less than 1% per year). Contraception should be continued for a period of 24 weeks after dosing has been completed.
* Ability to comply with treatment, procedures and pharmacokinetics (PK) sample collection and the required study follow-up procedures

Exclusion Criteria:

* Accepted any other anti-tumor drug therapies within 4 weeks before fist dose
* Accepted radiotherapy within 4 weeks before enrollment
* An anthracyclines antibiotic treatment was received exceeding 320 mg/m² or other equivalent dose antharcyclines
* Subjects are eligible with clinically controlled and stable neurologic function >= 4 weeks, which is no evidence of CNS disease progression; Subjects with spinal cord compression and cancerous meningitis are not eligible
* Subjects receiving immunosuppressive agents (such as steroids) for any reason should be tapered off these drugs before initiation of trial treatment (with the exception of subjects with adrenal insufficiency, who may continue corticosteroids at physiologic replacement doses, equivalent to < 10 mg prednisone daily, inhaled steroids and topical use of steroids)
* Vaccination within 28 days of the first administration of trial treatment, except for administration of inactivated vaccines (e.g., inactivated influenza vaccines)
* Pregnant or nursing females；or intend pregnancy within this study period or within 6 monthes after the end of this study
* Severe chronic and active infection, need to system antibiosis/antiviral treatment
* Has interstitial lung disease, or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management
* Cavity effusion (pleural effusion, ascites, pericardial effusion, etc.) are not well controlled, and need locally treatment or repeated drainage

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity（DLT） | 28 days
  Dose-limiting toxicity
Objective response rate (ORR) | up to 2 years
  Objective response rate (ORR) per RECIST 1.1 criteria according to investigators assessment
Duration of response (DOR) | up to 2 years
  Duration of response (DOR) per RECIST 1.1 criteria according to investigators assessment

SECONDARY OUTCOMES:
Clinical benefit rate | up to 2 years
  Clinical benefit rate
Progression free survival (PFS) rates | 6 months and 12 months
  Progression free survival (PFS) rates
Overall survival (OS) rates | 6 months and 12 months
  Overall survival (OS) rates

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD,PhD, Principal Investigator — Peking University
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No